CLINICAL TRIAL: NCT06536608
Title: The Effect of Oketani Breast Massage on Breastfeeding Success, Breastfeeding Self-Efficacy and Satisfaction in Primiparous Mothers: A Randomized Controlled Trial
Brief Title: The Effect of Oketani Breast Massage on Breastfeeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Filiz Ünal Toprak, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FÜT-02
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Breast Feeding; Massage
Keywords: Breast Feeding; Nursing; Massage
MeSH Terms: conditions — Breast Feeding | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Two groups with oketani massage group and control group
Who Masked: Participant
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Group (Experimental): Pregnant women who meet the inclusion criteria assigned to the Oketani Massage group will be informed about the study and their written and verbal consent will be obtained. Pregnant women will be asked to fill out the 'Introductory Characteristics Information Form' and 'Prenatal Breastfeeding Self-Efficacy Scale Short Form' at the first meeting before the training and then they will be given breastfeeding training and massage prepared with the Oketani method. 2 weeks after the training, the researcher will apply Oketani breast massage twice before the mother enters the operating room and once before the mother's first breastfeeding in the operating room or in the ward. One day after birth, they will be asked to answer the Postpartum Breastfeeding Self-Efficacy Scale Short Form, LACTH and Visual Comparison Scale Satisfaction (VAS-S) scale.
  Interventions: Other: Massage
- Control Group (No Intervention): Pregnant women who meet the inclusion criteria and who are assigned to the control group will be informed about the study and their written and verbal consent will be obtained. Pregnant women will be asked to fill out the 'Introductory Characteristics Information Form' and 'Prenatal Breastfeeding Self-Efficacy Scale Short Form' at the first meeting. One day after birth, they will be asked to answer the Postpartum Breastfeeding Self-Efficacy Scale Short Form and LACTH.

INTERVENTIONS:
Other: Massage — The Oketani Method is based upon practical breastfeeding theory, but is original in its practice. Oketani breast massage improves breastmilk secretion, can prevent and treat problems such as mastitis. In addition, the massage is painless, allowing your body to relax and breathe, something very much appreciated by mothers.
  The Oketani breast massage consists of massaging and milking the base of the breasts. These delicate glands are massaged as well as protected.
  Other Names: Oketani Massage
  Arms: Massage Group

SUMMARY:
This study aims to determine the effects of Oketani breast massage on breastfeeding success, breastfeeding self-efficacy and satisfaction of primiparous mothers.

DETAILED DESCRIPTION:
Breastfeeding is the most important factor in infant nutrition. Breast milk is a nutritional source that contains the necessary nutrients for the healthy growth of infants after birth and has many benefits in terms of growth and development. However, although the rate of breastfeeding has increased today compared to the past, it is still not at the desired level. In order to increase breastfeeding rates, breastfeeding trainings and massage should be given starting from the prenatal period. It is important for health professionals to provide training and consultancy to women in order to manage the breastfeeding process correctly, which is important for the health of both the mother and the baby. In this direction, as a result of this study, it is thought that correct breastfeeding behavior and self-sufficiency will be developed in mothers by using the oketani breast massage method. No study has been found in our country where this method is used. In this respect, the study is original. As a result of the study, it is thought that the use of oketani breast massage by health professionals while providing breastfeeding education and consultancy will facilitate the breastfeeding process.

ELIGIBILITY:
Inclusion Criteria:

* To volunteer to participate in the study,
* To be over 18 years of age,
* To be able to read and write,
* To be able to read and understand Turkish,
* To have no hearing, speech or visual impairments,
* To have received breastfeeding training at a pregnancy school,
* To be healthy in the 36th week of primiparous pregnancy.

Exclusion Criteria:

* Obstacles to communication include having a visual, hearing or perception disorder,
* Not being able to read or write,
* Having a psychiatric illness,
* Being multiparous and having a vaginal birth,
* Having a risky pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women 36 weeks and over
Enrollment: 60 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-05-04 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Antenatal and Pospartum Breastfeeding Self-Efficacy Scale Short Form | 1. week, 2. week and after labor 1. day
  The first form of the scale developed by Dennis and Faux was designed as 33 items, but after a second study, Dennis revised the scale and created a 14-item short form. The Turkish validity and reliability study of the scale was conducted by Aluş Tokat et al. in 2017. The scale can be administered in prenatal and postnatal periods and measures how competent women feel about breastfeeding. The items of the five-point Likert-type scale are scored as not at all sure
  (1), not very sure (2), sometimes sure (3), sure (4), very sure (5). The lowest score that can be obtained from all the evaluation scores of the scale is 14 and the highest score is 70. A low total score on the scale indicates a low perception of breastfeeding self-efficacy. In the original scale, the Cronbach's alpha reliability coefficient of the prenatal form was 0.87 and the Cronbach's alpha reliability coefficient of the postnatal form was 0.86.

SECONDARY OUTCOMES:
Visual Assessment Scale - Satisfaction (VAS - S) | After labor 1. day
  The VAS is also used to measure other components besides pain, such as satisfaction.In our study, the VAS will also be used to assess mothers' breastfeeding satisfaction levels. The Visual Assessment Scale - Satisfaction (VAS-S) is a 10 cm ruler with the expression "Not satisfied" on one end and "Very satisfied" on the other end. The mother is asked to rate her satisfaction with breastfeeding after the training from 1 to 10. High scores on the scale indicate that the satisfaction of the recipients is also high

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Ünal Toprak, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Cankiri State Hospital, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No